CLINICAL TRIAL: NCT00633776
Title: Perforomist Versus Foradil Evaluated by Inspiratory Capacity and HRCT
Brief Title: Perforomist Versus Foradil Evaluated by Inspiratory Capacity and High Resolution Computed Tomography (HRCT)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew funding prior to study initiation
Sponsor: University of California, Los Angeles (Other)
Collaborators: Dey, L.P. (Unknown)
Responsible Party: Donald Tashkin, M.D., University of California, Los Angeles (UCLA) David Geffen School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Perforomist CT Study
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Chronic Bronchitis; Emphysema
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Chronic bronchitis; Emphysema; Perforomist; Foradil; CT; lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Formoterol fumarate 20 mcg (Perforomist) nebulized via Pari C nebulizer at Test Visit 1; Formoterol 12 mcg (Foradil) via aerosolizer dry powder inhaler at Test Visit 2
  Interventions: Drug: formoterol fumarate
- 2 (Active Comparator): Formoterol fumarate 12 mcg (Foradil) via aerosolizer dry powder inhaler at Test Visit 1; Formoterol fumarate 20 mcg (Perforomist) nebulized via Pari C nebulizer at Test Visit 2
  Interventions: Drug: formoterol fumarate

INTERVENTIONS:
Drug: formoterol fumarate — Nebulized formoterol fumarate 20 mcg one-time treatment; aerosolizer dry powder formoterol fumarate 12 mcg one-time treatment
  Other Names: Perforomist (nebulized formoterol fumarate); Foradil (aerosolizer dry powder formoterol fumarate)

SUMMARY:
The purpose of this study is to compare the effects of nebulized formoterol fumarate (Perforomist) to dry-powder inhaler formoterol fumarate (Foradil). Perforomist is a solution that is made into very fine spray (using a nebulizer) that is then breathed in over 10-15 minutes. Foradil is taken in a single quick, deep inhalation.

DETAILED DESCRIPTION:
Participation requires 3 visits over 1-5 weeks. The first visit (Screening) will help determine subjects' eligibility through medical history, physical exam, lung function testing, and exercise testing. Those who qualify will be invited back to 2 test visits, at which subjects will undergo lung function testing and high-resolution CT scans before and after treatment with one of the study drugs. All subjects will take both study drugs: those who are randomized to Perforomist at Test Visit 1 will take Foradil at Test Visit 2, and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects with moderate to severe COPD
* Age greater than/equal to 40 years
* History of smoking greater than/equal to 20 pack-years of cigarettes
* No history of asthma (in the opinion of the investigator)
* No COPD exacerbations within the past 2 months requiring oral corticosteroids or hospitalization.
* No continuous oxygen therapy
* Subjects with a body mass index less than 15 or greater than 38
* Patients must be without other clinically significant illnesses or condition that might interfere with the study, including but not limited to uncontrolled hypertension, cardiovascular disease, cardiac arrhythmia, diabetes, hyperthyroidism, seizure disorder or any history of pheochromocytoma
* Be using medically acceptable birth-control measures if a female of child-bearing potential
* Not be pregnant or breastfeeding
* Be willing to withhold any existing short or long-acting bronchodilators for the appropriate time period prior to each test day (see below). Use of inhaled corticosteroids is not exclusionary, but will be maintained at a constant level throughout the study.
* Must be willing and able to perform spirometry, slow vital capacity, plethysmography, DLCO, and 6 minute walk after appropriate instruction.
* No known allergy or contradiction to albuterol or formoterol or prior significant adverse reactions to other beta agonists.
* No hypersensitivity to milk protein. Bloating or gas from lactose is not an exclusion.
* No use of beta-blockers (selective or non-selective), phenothiazines (thioridazine), or other drugs that may interact with formoterol or albuterol for the duration of the study. Washout of greater than seven half-lives of the drug prior to the study.
* No use of cardiac anti-arrhythmics Class Ia (e.g., disopyramide, procainamide, quinidine), or class III (e.g., amiodarone, dofetilide, ibutilide, sotalol), terfenadine, astemizole, mizolastine and any other drug with potential to significantly prolong the QT interval.
* No use of non-potassium sparing diuretics unless in fixed combination with potassium sparing diuretic.
* No investigational drugs within 30 days
* No subjects affiliated with the Division of Pulmonary, Critical Care Medicine and Hospitalists, David Geffen School of Medicine
* Informed consent

Exclusion Criteria:

* Post-albuterol FEV1/FVC less than lower limit of normal (Hankinson)
* Post-albuterol FEV1 between 30% and 60% predicted (Hankinson)
* An increase in FEV1 after albuterol sulfate HFA of at least 5% and 50 ml

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Distal airway measurements in COPD using inspiratory capacity as measure of small airways patency | End of study

SECONDARY OUTCOMES:
Differences in anatomic lobar air-trapping by HRCT due to small airways dilation between Perforomist and Foradil | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Donald P Tashkin, M.D., Principal Investigator — University of California, Los Angeles; Eric Kleerup, M.D., Study Director — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States